CLINICAL TRIAL: NCT05877677
Title: The Effects Assessment of the Polygonatum Kingianum Extract on Endurance Performance and Anti-fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-027-A
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator): consume 1 bottle per day
  Interventions: Dietary Supplement: Placebo drink
- Polygonatum kingianum extract drink (Experimental): consume 1 bottle per day
  Interventions: Dietary Supplement: Polygonatum kingianum extract drink

INTERVENTIONS:
Dietary Supplement: Placebo drink — consume 1 bottle per day
  Arms: Placebo drink
Dietary Supplement: Polygonatum kingianum extract drink — consume 1 bottle per day
  Other Names: Dragon Power® Polygonatum kingianum extract drink
  Arms: Polygonatum kingianum extract drink

SUMMARY:
To assess the efficacy of polygonatum kingianum extract on endurance performance and anti-fatigue

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 30-60 years old
* Must read and sign the informed consent form
* During the experiment, do not change the lifestyle and eating habits
* Cooperate not to engage in high-intensity exercise 48 hours before each experiment

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* People with serious diseases of heart, liver, kidney, endocrine and other organs (such as hypertension, diabetes, renal dysfunction and heart-related diseases) and mental patients
* People who have undergone surgery within 6 months or have lower limb injuries
* People who are allergic to Polygonatum kingianum extract
* Participate in other clinical trials related to anti-fatigue within four weeks of the trial
* Students who are currently taking courses taught by the principal investigator of this trial.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The change of aerobic endurance | Day 0, day 14, day28
  3-min step test is used to assess aerobic endurance
The change of continuous attention performance | Day 0, day 14, day28
  Canon continuous attention software (Conners' Continuous Performance Test) is used to assess continuous attention performance
The change of concentration of testosterone in blood | Day 0, day 14, day28
  Fasting venous blood was sampled to measure concentrations of testosterone
The change of blood PDE5 gene expression | Day 0, day 14, day28
  Fasting venous blood was sampled to measure the expression of PDE5 gene

SECONDARY OUTCOMES:
The change of blood nitric oxide (NO) | Day 0, day 14, day28
  Fasting venous blood was sampled to measure concentrations of nitric oxide
The change of self-assessment fatigue condition | Day 0, day 14, day28
  A 10 point likert scale was utilized to evaluate fatigue condition. The higher the score, the higher the fatigue level.

OTHER OUTCOMES:
The change of concentrations of liver function biomarkers (AST, ALT) in blood | Day 0, day 14, day28
  Fasting venous blood was sampled to measure the concentration of liver function biomarkers- Aspartate amino transferase (AST), Alanine amino transferase (ALT).
The change of concentrations of renal function biomarkers (BUN, creatinine) in blood | Day 0, day 14, day28
  Fasting venous blood was sampled to measure the concentration of renal function biomarkers- Blood Urea Nitrogen (BUN), creatinine.
The change of concentrations of blood lipid profiles (total cholesterol, LDL-C, HDL-C, triglyceride) | Day 0, day 14, day28
  Fasting venous blood was sampled to measure lipid profiles- total cholesterol, Low Density Lipoprotein-Cholesterol (LDL-C), High Density Lipoprotein-Cholesterol (HDL-C), triglyceride.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-han Wu, Principal Investigator — National Pingtung University of Science and Technology
Locations (1):
- National Pingtung University of Science and Technology, Pingtung City, Taiwan